CLINICAL TRIAL: NCT03242070
Title: A Theory-Based Patient Portal eLearning Program for Older Adults With Chronic Illnesses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Eun-Shim Nahm, Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HP-00069040
Record Dates: First submitted 2017-08-02; First posted 2017-08-08 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Patient Portals; Chronic Disease; Older Adults
Keywords: Patient Portals; Chronic Disease; Older Adults
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Intervention Model Description: A two-arm parallel-group RCT
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Theory-based PP eLearning Program(T-PeP) (Experimental): Theory-based PP eLearning Program (T-PeP) was developed based on self-efficacy theory42-44 to improve older adults' use of PPs for managing their care and includes learning modules, discussion boards, and other resources. Considering variations in the types and usability of PPs used by patients nationwide, T-PeP was developed as a vendor-agnostic ("not tied to a specific vendor") program.
  Interventions: Other: Theory-based PP eLearning Program(T-PeP)
- Control Group (No Intervention): No specific intervention will be provided to the control group participants

INTERVENTIONS:
Other: Theory-based PP eLearning Program(T-PeP) — Theory-based PP eLearning Program (T-PeP) was developed based on self-efficacy theory42-44 to improve older adults' use of PPs for managing their care and includes learning modules, discussion boards, and other resources. Considering variations in the types and usability of PPs used by patients nationwide, T-PeP was developed as a vendor-agnostic ("not tied to a specific vendor") program.
  Arms: Theory-based PP eLearning Program(T-PeP)

SUMMARY:
The high prevalence of chronic illnesses is a serious public health problem in the U.S., and more than 70 million adults age ≥50 have at least one chronic illness. Management of chronic conditions requires long-term use of complex treatment plans and can cause unintended consequences, such as increased risk of medication errors. Patient portals (PPs), a federally supported health information technology (IT), can be especially helpful for patients with chronic illnesses. Patients can now access their own health records and directly communicate with care providers through PPs. Prior findings suggest a great potential for using PPs to improve care quality, and the federal government funds healthcare organizations to implement this tool nationwide. Despite the potential benefits, the overall PP adoption rate in the U.S. is low. A lack of PP use among older adults has been addressed as a particular concern. When only older adults who use the Internet are considered, however, their proportion of PP use is similar to other age groups. A few studies also reported that older adults are receptive to PPs. In general, older adults need additional support for learning to use PPs, as they tend to be less familiar with technology. Currently, most older adults receive little or no PP support from their providers. This is an important gap in the nation's health IT initiative because without appropriate support, older adults will not be able to use this robust health tool, missing an important opportunity to improve their health outcomes. In an effort to fill this gap, the investigators developed and tested an older adult friendly Theory-based Patient portal eLearning Program (T-PeP) to support older adults in using PPs for their care. In the proposed feasibility study, the investigators plan to (Aim 1) optimize and implement a vendor-agnostic T-PeP and conduct formative and process evaluations; and (Aim 2) assess the preliminary impact of T-PeP on PP use and selected outcomes (PP knowledge, self-efficacy for PP use and health decision making, health communication, and medication reconciliation). If successful, this study could directly affect quality of care provided to older adults and the success of the national health IT initiative. Findings from this study will also provide hospitals, vendors, and policymakers with in-depth information on older adults' current PP usage patterns and other challenges in using various types of PPs at the national level.

DETAILED DESCRIPTION:
The high prevalence of chronic illnesses is a serious public health problem in the United States, accounting for 70% of all deaths. Older adults are especially vulnerable; more than 70 million adults age ≥50 have at least one chronic illness (e.g., heart disease, diabetes). Management of chronic conditions requires long-term use of multiple medications and complex treatment plans, which can cause unintended consequences, such as increased risk of medication errors. Engaging patients in their care and health decision-making processes is vital for the provision of high quality care to people with chronic conditions. Until recently, however, patients were not given access to their own health records and had to call their providers' offices to communicate with them. In the past few years, the nation has made unprecedented efforts to transform health care using information technology (IT). Through secure patient portals (PPs), patients now can access their electronic health records (EHRs), directly send eMessages to their providers, and request medication renewals online. They can also involve their family caregivers in their care more efficiently. PPs are especially helpful for patients with chronic illnesses, as they offer tools to manage health conditions. With the Meaningful Use (MU) incentive payment program by the Centers for Medicare and Medicaid Services (CMS), healthcare organizations nationwide are implementing PPs and making them available to the public.

Prior findings demonstrated positive impacts of PPs on management of chronic conditions, adherence to treatment, and patient-provider communication. Currently, PP adoption rates vary depending on care organizations, but the overall nationwide adoption rate has been low (26.8%). A lack of PP use among older adults has been addressed as a particular concern. Based on 2014 national survey data, however, when only online users were considered, the proportion of PP use in older adults was similar to other age groups (≥18 yrs, 32.2%; 50-64, 34.1%; ≥65, 29.8%). In a 2015 SeniorNet34 member survey (N=553; mean age, 73.6 yrs), 60.6% (n=327) reported having at least one PP account. These findings indicate an excellent potential for using PPs for the care of older adults (AHRQ's priority population36). Many older adults, however, are not technologically savvy and need additional support. Currently, most older adults receive little or no PP training support from their providers. This is a critical gap in the nation's health IT initiative because without appropriate support, older adults will not be able to use this robust health tool, missing an important opportunity to improve their health-related outcomes.

In an effort to fill this gap, in our previous studies the investigators developed and tested the older adult friendly Theory-based PP eLearning Program (T-PeP) to provide older adults necessary support for using PPs. In the proposed feasibility study, the investigators will optimize and implement the program in a large older adult online community, conduct formative/process evaluation, and assess its preliminary impact on PP use and selected health-related outcomes. T-PeP was developed based on self-efficacy theory to improve older adults' use of PPs for managing their care and includes learning modules, discussion boards, and other resources. Considering variations in the types and usability of PPs used by patients nationwide, T-PeP was developed as a vendor-agnostic ("not tied to a specific vendor") program. The specific aims of the study are to:

Aim 1: Optimize and implement T-PeP in an older adult online community and conduct formative and process evaluations (e.g., usability problems, barriers and facilitators for PP use, and other practical issues).

Aim 2: Assess the preliminary impact of T-PeP on older adults' PP use and selected health-related outcomes using a two-arm randomized controlled trial (RCT). Older adult online users with chronic conditions (N=242, age ≥50) will be recruited from a large older adult online community (SeniorNet.org).

H1. The intervention group participants will demonstrate greater improvement than the control group at the end of T-PeP (3 weeks) and at 4 months in PP knowledge, self-efficacy for using PPs and making health decisions, perceived patient-provider communication, and PP use (enrollment, usage frequency).

H2. More participants in the intervention group than the control group will reconcile the medications they are taking with the medications listed in their PP at 4 months.

This study could directly impact quality of care provided to older adults and the success of a national health IT initiative by offering a critically missing component in the current PP implementation process-patient support for the health IT (PP) designed for patients. Findings from the study will also provide hospitals, vendors, and policymakers in-depth information on older adults' current PP usage patterns and other challenges in using various PPs at the national level, contributing to the improvement of PP technology and clinical practices. Once the feasibility of the study is demonstrated, the vendor-agnostic T-PeP could be used widely and incorporated into busy practices. The next R01 study will test its long-term effects on health behavior and clinical outcomes, as well as care cost, using more diverse samples, including practice settings and underserved populations.

ELIGIBILITY:
Inclusion Criteria:

* being age ≥50
* having been diagnosed with at least one chronic disease* (e.g., heart disease, diabetes, cancer)
* having access to the Internet/e-mail
* being able to use the Internet/e-mail independently
* currently residing in the U.S.
* being able to read/write English.

Exclusion Criteria:

-

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 276 (Estimated)
Dates: Start 2017-01-17 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
PP knowledge | Change from baseline knowledge at 3 week and 4 months
  An 8-item questionnaire developed by experts and tested in preliminary studies (α=.50).40,41
Self-efficacy for using PPs | Change from baseline knowledge at 3 week and 4 months
  a modified 4-item Self-Efficacy for Computer-Based PHR Scale100 (α=.97; criterion validity), which was successfully used in our preliminary studies.40,41
Self-efficacy for health decision making | Change from baseline knowledge at 3 week and 4 months
  Decision Self-Efficacy Scale, including 11 items on a 5-point Likert scale. The scale assesses the person's ability to obtain information, ask questions, and make a choice.136-138 It was tested for older adults in an eHealth study (α=.83; criterion validity).139
Patient-provider communication | Change from baseline knowledge at 3 week and 4 months
  14 items of the Components of Primary Care Instrument140,141 that assesses the following 3 areas: interpersonal communication, physician's knowledge of the patient, coordination of care. This tool has been tested in our prior study40 (α=.89; factor analysis141).
PP use | Change from baseline knowledge at 3 week and 4 months
  The number of newly activated account(s) and the frequency of PP usage per function; lab results, medications, and health summaries; and other functions as reported in the scheduled surveys.

SECONDARY OUTCOMES:
Medication reconciliation | Change from baseline knowledge at 3 week and 4 months
  The frequency of comparing all medications that participants are taking with all medications listed on their PP142 as reported in the scheduled surveys.

CONTACTS AND LOCATIONS:
Locations (1):
- SeniorNet, Fort Myers, Florida, United States

IPD SHARING:
Plan to Share IPD: No